CLINICAL TRIAL: NCT01729507
Title: Transcranial Direct Current Stimulation (TDCS) as Add on Therapy for Treatment of Tobacco Dependence by Standardized Behaviour Therapy - Active and Placebo Controlled Double Blind Study
Brief Title: tDCS as Add on Therapy for Treatment of Tobacco Dependence by Standardized Behaviour Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Andrea Linhardt, physician, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 489-11
Record Dates: First submitted 2012-05-28; First posted 2012-11-20 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Smoking Cessation; Tobacco Dependence
Keywords: Smoking cessation; Add on and smoking cessation; Therapy for tobacco dependence; Transcranial direct current stimulation
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment with tDCS (Active Comparator): This group will receive 7x verum treatment with tDSC. All participants receive standardised behavioural therapy ('The smoke-free programme')
  Interventions: Other: tDCS; Behavioral: standardised behavioural therapy
- 7x sham treatment (Placebo Comparator): This group will receive 7x sham treatment. All participants will receive standardised behavioural therapy ('The smoke-free programme')
  Interventions: Behavioral: standardised behavioural therapy

INTERVENTIONS:
Other: tDCS — Stimulation will be performed with a DC stimulator MC Location of stimulation: Anode over the left dorsolateral cortex, corresponding with F3 (in 10-20 EEG system); cathode over the right temporal cortex Intensity: 2 mA Total duration: Constant stimulation for 20 minutes
  Other Names: Stimulator MC (neuroConn GmbH, Ilmenau, Germany).
  Arms: Treatment with tDCS
Behavioral: standardised behavioural therapy — The standardised behavioural therapy will be performed according to the certified "Smoke-free programme' of the of the Institute for Therapy Research ('Institut für Therapieforschung', IFT). The course leaders' manual specifies that the ideal number of participants is 8-12.
  1 group session for 90 minutes/week for 7 weeks, 2 telephone calls of 10 minutes each, first after the fourth session 3 days after collective smoking cessation, second on day 3 after the last session.

SUMMARY:
As an add-on treatment to behavioural therapy for tobacco dependence, anodal transcranial direct current stimulation (tDCS) significantly increases the cessation rate compared to treatment with sham tDCS; endpoint analysis will be performed 1, 3, 6 and 12 months after completion of the smoke-free programme in combination with tDCS.

Craving, assessed with a visual analog scale (VAS), is reduced significantly in the verum treatment group compared to the sham tDCS group.

tDCS is suitable for use in larger groups (8-12 people).

DETAILED DESCRIPTION:
1. General design and study population

   Controlled, randomised, double-blind study with no crossover; sample size estimate: 20-36 participants.

   Sample size calculations are not necessary for pilot studies. A general 'rule of thumb' is to use 30 or more patients.

   An interim analysis of the data will be performed after completion of the second course (stimulation of 24 patients). We reserve the right to increase the sample size by 12-24, depending on the effect size, so that we have data from 30 participants per arm and the estimate is reliable.

   Study participants will be recruited via newspaper advertisements, advertisements on the internet page of the tobacco outpatient clinic and announcements on notice boards in the Department of Psychiatry.

   Study duration: it is estimated that 12 days will be required for each patient to complete the study protocol. The total study duration for 36 patients is estimated to be 12 months.
2. Screening

   No screening investigations will be performed.
3. Randomisation and blinding

   Patients will be randomised to two groups of 10-18 patients each. One group will receive 7x verum treatment with tDSC, the other 7x sham treatment. All participants will then receive standardised behavioural therapy ('The smoke-free programme'). Both patients and clinical raters will be blind to the treatment condition. Unblinding will take place only after completion of the study or if the whole study is discontinued because of severe incidents.
4. Experimental paradigm

   Up to 12 participants (maximum number of participants for the smoke-free programme) will be stimulated per course. A total of 3x12 participants will be stimulated during the study and subsequently participate in the certified behavioural therapy 'Smoke-free programme' by Gradl, S. and Kröger, C. (2008).

   Blinding will be performed before the start of the study. Every participant will be given a number (pseudonym), which will be programmed into the stimulator. Each number will be randomly assigned to sham or verum treatment and the same treatment will then be performed at every session. The stimulator can be programmed beforehand to assign numbers randomly to the verum or sham group, so that the respective patient data are unknown to both the person who performs the stimulation and the course leaders. Half of the participants will be randomly assigned to the sham group and half to the verum group. The stimulator will be programmed at the start of the study.

   Stimulation will be performed with a DC stimulator MC (neuroConn GmbH, Ilmenau, Germany). The stimulator is a micro-processor-controlled constant current source with up to 16 freely programmable independent channels. The maximum current strength is 5 mA and the maximum stimulation duration 30 minutes. The stimulator is a CE-certified medical product that has been used in various national and international studies.

   The current is transmitted via sponge electrodes (35 cm2) soaked in physiological salt solution. The electrodes are attached to the head with elasticated bands.

   Location of stimulation: Anode over the left dorsolateral cortex, corresponding with F3 (in 10-20 EEG system); cathode over the right temporal cortex; Intensity: 2 mA; Total duration: Constant stimulation for 20 minutes, plus 15 seconds ramp-in and ramp-out phase during which the current will be regulated up and down, respectively.

   Stimulation time schedule: Each participant will be stimulated a total of 7 times over 7 weeks.

   The stimulation will be followed by a 90-minute session of the 'Smoke-free programme'.

   The standardised behavioural therapy will be performed according to the certified "Smoke-free programme' of the of the Institute for Therapy Research ('Institut für Therapieforschung', IFT). The course leaders' manual specifies that the ideal number of participants is 8-12.

   IFT 6-week course

   Schedule:

   Duration: 7 weeks 1 group session for 90 minutes/week for 7 weeks 2 telephone calls of 10 minutes each, first after the fourth session 3 days after collective smoking cessation, second on day 3 after the last session.

   Study procedures:
   * 1st session: Smoking and a smoke-free life
   * 2nd session: The smoker's ambivalence
   * 3rd session: Errors in reasoning and alternatives
   * 4th session: Preparing to quit smoking

   SMOKING CESSATION
   * 1st telephone call: Individual telephone support
   * 5th session: Experiences from quitting smoking
   * 6th session: Identity as a smoke-free person
   * 7th session: Planning the future
   * 2nd telephone call: Individual telephone support
5. Evaluation scales

   * Edinburgh Handedness Test: Test to assess left- or right-handedness to evaluate the dominant hemisphere.
   * Comfort Rating Questionnaire: Questionnaire to record symptoms after tDCS
   * Fagerström Test: Questionnaire to evaluate physical tobacco dependence
   * Questionnaire on Smoking Urges (Tiffany & Drobes, 1991) (German version: Müller, Mucha, Ackermann & Pauli, 2001): Uses two scales to measure craving for cigarettes.
6. Additional evaluations

   As an additional evaluation, at the start of the stimulation and at four follow-up appointments salivary cotinine (a degradation product of tobacco) and the carbon monoxide content of expired air will be measured. Carbon monoxide will be measured with a Micro Smokerlyzer (Bedfont Scientific Ltd., Maidstone, England).

   At the end of each tDCS treatment, the study participants will complete a Comfort Rating Questionnaire (CRQ). Our research group has used this questionnaire about direct current stimulation for several years and has continually improved and updated it. The questionnaire records unpleasant sensations and side effects during and after direct current stimulation.
7. Sample size estimate

   Sample size estimation and study design correspond with the usual procedures in comparable pilot studies (e.g. on tDCS or TMS).
8. Statistical analysis

Data will be analysed with a multivariate analysis of covariance (MANCOVA). The absolute values of the evaluation scales will be the dependent variables and the treatment condition the independent factor.

ELIGIBILITY:
Inclusion criteria:

* Age of legal majority
* Smoker for > 1 year, >10 cigarettes/day
* CO>10ppm; measurement in expired air by means of a Micro Smokerlyzer (Bedfont Scientific Ltd., Maidstone, England)
* Quantification of tobacco dependence with the Fagerström Test
* The patient should not have attempted to quit smoking or have received drug treatment for quitting smoking for at least 3 months before the start of the study
* Ability to give informed consent

Exclusion Criteria:

* Acute psychiatric disorders according to ISD-10/DSM-IV
* Under legal care
* Pregnancy
* Contraceptive methods with a Pearl Index >1
* Other severe psychiatric disorders
* Acute suicidality
* Drug, medication or alcohol abuse at the time of the study
* Dementia (DSM-IV/ICD-10 criteria)
* History of severe craniocerebral trauma
* Indications of structural damage to the basal ganglia or the brain stem
* Severe neurological disorders (such as prolapsed disk in the past 6 months, polyneuropathy, Parkinson syndrome, epilepsy, dementia, systemic neurological diseases, cerebrovascular diseases, history of stroke, repeated cerebral ischaemia with progressive worsening, elevated cerebral pressure, normal pressure hydrocephalus)
* Severe medical disorders (such as manifest arterial hypertension, severe cardiovascular disorders, cardiac pacemaker, respiratory insufficiency)
* Any electronic implants
* Malignant diseases of any kind, also in the medical history
* Severe active infectious diseases
* Chronic and systemic skin diseases
* Bone diseases (such as Paget's disease, osteoporosis with spontaneous fractures, fresh fractures)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
cessation rate | at 4 weeks after last intervention
  salivary cotinine in ng/ml and the carbon monoxide content of expired air (COppm and %COHb)will be measured.

SECONDARY OUTCOMES:
Craving | week one directly before first tDCS intervention
  Craving, assessed with a visual analog scale (VAS)and Questionnaire on Smoking Urges (QSU), is reduced significantly in the verum treatment group compared to the sham tDCS group.
Craving | week two directly before second tDCS intervention
  Craving, assessed with a visual analog scale (VAS)and Questionnaire on Smoking Urges (QSU), is reduced significantly in the verum treatment group compared to the sham tDCS group.
Craving | week three directly before third tDCS intervention
  Craving, assessed with a visual analog scale (VAS)and Questionnaire on Smoking Urges (QSU), is reduced significantly in the verum treatment group compared to the sham tDCS group.
Craving | week four directly before fourth tDCS intervention
  Craving, assessed with a visual analog scale (VAS)and Questionnaire on Smoking Urges (QSU), is reduced significantly in the verum treatment group compared to the sham tDCS group.
Craving | week five directly before fifth tDCS intervention
  Craving, assessed with a visual analog scale (VAS)and Questionnaire on Smoking Urges (QSU), is reduced significantly in the verum treatment group compared to the sham tDCS group.
Craving | week six directly before sixth tDCS intervention
  Craving, assessed with a visual analog scale (VAS)and Questionnaire on Smoking Urges (QSU), is reduced significantly in the verum treatment group compared to the sham tDCS group.
Craving | week seven directly before seventh tDCS intervention
  Craving, assessed with a visual analog scale (VAS)and Questionnaire on Smoking Urges (QSU), is reduced significantly in the verum treatment group compared to the sham tDCS group.
Craving | four weeks after last intervention
  Craving, assessed with a visual analog scale (VAS)and Questionnaire on Smoking Urges (QSU), is reduced significantly in the verum treatment group compared to the sham tDCS group.
Craving | twelve weeks after last intervention
  Craving, assessed with a visual analog scale (VAS)and Questionnaire on Smoking Urges (QSU), is reduced significantly in the verum treatment group compared to the sham tDCS group.

OTHER OUTCOMES:
cessation rate | at 12 weeks after last intervention
  salivary cotinine in ng/ml and the carbon monoxide content of expired air (COppm and %COHb)will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Padberg, PD Dr., Study Director — Department of Psychotherapy and Psychosomatic Medicine
Locations (1):
- Ludwig Maximilans University, Munich, Bavaria, Germany